CLINICAL TRIAL: NCT01276275
Title: A Pharmacoepidemiological Study to Examine Patient Characteristics, Drug Utilization Pattern and Crude Incidence Rates of Selected Outcomes in New Users of Ticagrelor, Clopidogrel and Prasugrel in National Swedish Registries
Brief Title: Extended Drug Utilization Study Among Patients Exposed to Ticagrelor, Clopidogrel and Prasugrel
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130N00010
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Bleeding ,Arrhythmias, Heart Failure, Acute Renal Failure, Acute Liver Failure, Dyspnoea, Gout
Keywords: Acute coronary syndrome, thienopyridine, epidemiology
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury; Liver Failure, Acute; Dyspnea; Gout; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exposure Group 1: First time users of ticagrelor
  Interventions: Drug: Risk of selected safety events
- Exposure Group 2: First time users of clopidogrel
  Interventions: Drug: Risk of selected safety events
- Exposure Group 3: First time users of prasugrel
  Interventions: Drug: Risk of selected safety events

INTERVENTIONS:
Drug: Risk of selected safety events — First time users of ticagrelor, clopidogrel and prasugrel, respectively

SUMMARY:
The purpose of the study is to describe patient characteristics and drug usage among patients that are prescribed ticagrelor for the first time and to compare them with patients who are prescribed clopidogrel and prasugrel for the first time.

A further purpose is to ascertain and estimate the crude incidence rate of bleeding, arrhythmias, heart failure, acute renal failure, acute liver failure, dyspnoea and gout among new users in the three cohorts of ticagrelor, clopidogrel and prasugrel.

ELIGIBILITY:
Inclusion Criteria:

* First time users of ticagrelor, clopidogrel and prasugrel, respectively

Exclusion Criteria:

* Individuals with more than one of above three antiplatelet drugs dispensed the same day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 20 to 84 years before their first study drug dispension (start date) will be included in the study. The study period will start the first month after ticagrelor market introduction in Sweden (the first of June 2011),
Sampling Method: Non-Probability Sample
Enrollment: 7200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Drug utilization: Description of patient characteristics and drug usage | Up to one year after entry into study cohort

SECONDARY OUTCOMES:
Follow-up of safety outcomes: First occurrence of bleeding, arrhythmias, heart failure, acute renal failure, acute liver failure, dyspnoea and gout | Up to one year after entry into study cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Kieler, MD, PhD, Assoc Prof, Principal Investigator — Centre for Pharmacoepidemiology, Karolinska Institute, Stockholm
Locations (1):
- Research Site, Stockholm, Sweden

REFERENCES:
- See also: SynopsisD5130N0010 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=488&filename=SynopsisD5130N0010.pdf